CLINICAL TRIAL: NCT01008319
Title: Traditional Clomiphene Citrate Administration Versus a Stair-Step Approach: A Randomized Controlled Trial
Brief Title: Traditional Clomiphene Citrate Administration vs. Stair-step Approach
Acronym: Clomid
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2078
Record Dates: First submitted 2009-11-03; First posted 2009-11-05 (Estimated); Results first posted 2018-01-08 (Actual); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: Ovulatory Dysfunction; Anovulation; Ovulation Induction
Keywords: Anovulation; Ovulation induction
MeSH Terms: conditions — Anovulation | interventions — Clomiphene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Traditional Administration (Active Comparator): The traditional approach to ovulation induction with clomiphene citrate involves administration of 50mg/day for five days (starting on cycle day 3, 4, or 5). If ovulation does not occur then a progestin is prescribed to induce menses (which occurs within one week of stopping the progestin) and then a higher dose of medication is used in the next cycle.
  Interventions: Drug: clomiphene citrate
- Stair-Step Administration (Experimental): The stair-step protocol the dose of clomiphene citrate would be increased without administering progestin and inducing a period. This would eliminate the days of progestin (10 days) and the waiting for the period (usually 3 to 7 days) and finally waiting to start clomiphene citrate on cycle day 3 at the earliest (3 more days) for a total of up to 20 days difference for the 100 mg dose of clomid. If they did not ovulate on 100mg, then the process repeats and another 20 days before they start 150mg. Therefore, the time to ovulation and pregnancy may be reduced, and hopefully pregnancy, by using the stair-step protocol. This method utilizes ultrasound monitoring for follicle development before increasing the dose of clomiphene citrate.
  Interventions: Drug: clomiphene citrate

INTERVENTIONS:
Drug: clomiphene citrate — Clomiphene citrate 50 mg for 5 days starting on cycle day 5. Transvaginal ultrasound between cycle days 11 to 14 to determine if there is a dominant follicle. If NO dominant follicle present, another ultrasound and blood draw (to test progesterone level) will be done one week later to confirm no response to the medication dose. Medroxyprogesterone acetate (Provera) 10 mg per day for 10 days. Increased dose of clomiphene citrate for 5 days starting on cycle day 5. This process will be repeated at increased doses of clomiphene citrate (100 mg and 150 mg) until a dominant follicle(s) is present.
  Other Names: Clomid
  Arms: Traditional Administration
Drug: clomiphene citrate — Clomiphene citrate 50 mg for 5 days starting on cycle day 5. Transvaginal ultrasound between cycle days 11 to 14 to determine if there is a dominant follicle. If NO dominant follicle present, a blood draw (to test progesterone level) will be done. Increased dose of clomiphene citrate for 5 days starting that day. A repeat transvaginal ultrasound in one week to determine if there is a dominant follicle. This process will be repeated at increased doses of clomiphene citrate (100 mg and 150 mg) until a dominant follicle(s) is present.
  Other Names: Clomid
  Arms: Stair-Step Administration

SUMMARY:
The purpose of this study is to compare the length of time to achieve ovulation and pregnancy with a traditional protocol administration of clomiphene citrate versus a stair step administration.

Our hypothesis is by using a stair-step approach in which a period is not induced between administrations of escalating doses of clomiphene citrate, the time to ovulation and pregnancy may be reduced.

DETAILED DESCRIPTION:
The traditional administration of clomiphene citrate for ovulation induction involves taking clomiphene citrate for 5 days. If ovulation does not occur within 14 days, a progestin pill (such as Provera) is prescribed for 10 days to induce a period (which normally occurs within 1 week of stopping the pill). Then a higher dose of clomiphene citrate will be prescribed.

The stair-step administration of clomiphene citrate for ovulation induction also involves taking clomiphene citrate for 5 days. In contrast, if ovulation does not occur within 7-9 days, a progestin pill (such as Provera) would NOT be taken to induce a period. The dose of clomiphene will then be increased. Therefore, this would do away with the 10 days of taking the progestin pill, and also do away with waiting for a period (usually 3 to 7 days) for a total of up to a 20 day difference between clomiphene citrate dosing cycles.

ELIGIBILITY:
Inclusion Criteria:

* Ovulatory dysfunction as evidenced by mid-luteal progesterone less then 3ng/dL, non-biphasic basal body temperature charting, or menstrual history of cycles > 35 days.
* Female patients 18 to 45 years old
* Six months or greater of unprotected intercourse without pregnancy.
* Normal TSH and prolactin serum levels
* Semen analysis of male partner with > 15 million motile sperm on semen analysis.

  * NOTE: Must be willing to travel to the Oklahoma City area for treatment.

Exclusion Criteria:

* Failure to spontaneously menstruate or to menstruate following progestin administration
* Allergy or intolerance to the side effects of clomiphene citrate, hCG (human chorionic gonadotropins), or medroxyprogesterone acetate (Provera).
* Known anatomical defect affecting the uterine cavity including submucosal fibroids or endometrial polyps.
* Know tubal hydrosalpinx or risk factors for tubal obstruction
* Known liver dysfunction
* Known or suspected androgen secreting tumor, cushings disease, or adrenal hyperplasia (congenital or adult onset)
* Ovarian cyst > 20mm or endometrial lining >6 mm on trans-vaginal baseline ultrasound.
* Stage III or IV endometriosis
* Decreased ovarian reserve as evidenced by antral follicle count less than 6 by Transvaginal ultrasound or a cycle-day-3 serum FSH of > 10 uIU/ml.
* Positive HIV in either the female patient or her partner.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2009-10; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: LaTasha Craig, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was in the infertility clinic.
Groups:
- Traditional Administration: The traditional approach to ovulation induction with clomiphene citrate involves administration of 50mg/day for five days (starting on cycle day 5). If ovulation does not occur by day 21 then a progestin is prescribed to induce menses (which occurs within one week of stopping the progestin) and then a higher dose of medication is used in the next cycle.
  This process will be repeated at increased doses of clomiphene citrate (100 mg and 150 mg).
- Stair-Step Administration: The stair-step protocol the dose of clomiphene citrate would be increased without administering progestin and inducing a period. This method utilizes ultrasound monitoring for follicle development before increasing the dose of clomiphene citrate.
Period: Overall Study
Arm/Group | Traditional Administration | Stair-Step Administration
Started | 60 | 60
Completed | 60 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: A total of 120 patients (60 stair-step, 60 traditional) were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Traditional Administration | Stair-Step Administration | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.88 (4.95) | 29.37 (3.96) | 28.65 (4.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 60 | 120
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 0 | 4
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 3 | 9
  White | 46 | 55 | 101
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to Ovulation With Each Protocol
Description: We hypothesized that time to ovulation would be shorter with stair-step protocol vs. traditional.
Time Frame: 5 years
Measure: Mean (Standard Error); unit: days
Arm/Group | Traditional Administration | Stair-Step Administration
Number analyzed (Participants) | 60 | 60
days | 31.1 (3.5) | 21.5 (0.9)

2. Secondary Outcome: Rate of Ovulation
Description: Rate of ovulation with each dose of clomid within each protocol
Time Frame: 5 years
Population: Proportion of subjects that ovulated at each dose of Clomid based on which protocol they were randomized to.
Measure: Count of Participants; unit: Participants
Groups:
- Traditional Protocol: The proportion that ovulated at the dose of Clomid of 60 patients in the traditional protocol.
- Stair-Step Protocol: The proportion that ovulated at the dose of Clomid of 60 patients in the stair-step protocol.
Arm/Group | Traditional Protocol | Stair-Step Protocol
Number analyzed (Participants) | 60 | 60
Participants
  Clomid 50mg | 45 | 26
  Clomid 100mg | 7 | 18
  Clomid 150mg | 1 | 10
  Clomid No Response | 7 | 6

3. Secondary Outcome: Delivery Outcomes
Description: Proportion of participants that delivered a baby based on which protocol they were randomized to.
Time Frame: 5 years
Population: Number of participants randomized to each arm.
Measure: Count of Participants; unit: Participants
Groups:
- Traditional Protocol: Proportion of subjects that delivered in the traditional protocol.
- Stair-Step Protocol: Proportion of subjects that delivered in the stair-step protocol.
Arm/Group | Traditional Protocol | Stair-Step Protocol
Number analyzed (Participants) | 60 | 60
Participants | 21 | 21

ADVERSE EVENTS:
Description: Questionnaire were administered at each appointment for ultrasound evaluation. They assessed none, mild, moderate or severe symptoms including: hot flashes, mood swings, breast tenderness, pelvic discomfort, nausea, vomiting, blurry vision, light sensitivity, headache, decreased urination, weight gain, insomnia, nervousness and leg pain.
Arm/Group | Traditional Administration | Stair-Step Administration
Serious Adverse Events (participants affected / at risk) | 2/60 | 3/60
Other Adverse Events (participants affected / at risk) | 60/60 | 60/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Traditional Administration (N=60) | Stair-Step Administration (N=60)
Birth Defect (Congenital, familial and genetic disorders) | 0 (0) | 2 (2)
Blurry Vision/Double Vision (Eye disorders) | 1 (1) | 1 (1)
Gallstones (Hepatobiliary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Traditional Administration (N=60) | Stair-Step Administration (N=60)
Vasomotor Flushes (hot flashes) (Endocrine disorders) | 32 (146) | 30 (83) — Hot Flashes
Mood Swings (Psychiatric disorders) | 32 (104) | 27 (67) — mood irritability
Breast tenderness (Reproductive system and breast disorders) | 21 (35) | 21 (30)
Pelvic Discomfort (Reproductive system and breast disorders) | 29 (75) | 18 (36)
Nausea (Gastrointestinal disorders) | 26 (48) | 15 (28)
Blurry Vision/Double Vision (Eye disorders) | 6 (9) | 3 (3)
Light sensitivity (Eye disorders) | 7 (19) | 1 (2)
Headaches (Nervous system disorders) | 34 (90) | 27 (53)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Decreased urination frequency (Renal and urinary disorders) | 0 (0) | 1 (1)
Weight gain (Endocrine disorders) | 11 (21) | 6 (9)
Insomnia (General disorders) | 15 (33) | 7 (13)
Nervousness (Psychiatric disorders) | 12 (21) | 3 (4)
Leg pain/leg swelling (Musculoskeletal and connective tissue disorders) | 4 (6) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes